CLINICAL TRIAL: NCT02392377
Title: Pilot Study of Correlation Between Molecular Phenotype and Response to Two Independent Treatment Regimens, Carboplatin and Paclitaxel vs. 5-Fluorouracil and Oxaliplatin Chemotherapy in Patients With Localized Esophageal Adenocarcinoma
Brief Title: Molecular Phenotyping in Predicting Response in Patients With Stage IB-III Esophageal Cancer Receiving Combination Chemotherapy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CASE9314; NCI-2015-00034 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CASE 9314 (Other: Case Comprehensive Cancer Center); K12CA076917 (NIH); P50CA150964 (NIH); P30CA043703 (NIH)
Record Dates: First submitted 2015-03-13; First posted 2015-03-19 (Estimated); Results first posted 2018-02-13 (Actual); Last update posted 2018-02-13 (Actual); Status verified 2018-01

CONDITIONS: Stage IB Esophageal Adenocarcinoma; Stage IIA Esophageal Adenocarcinoma; Stage IIB Esophageal Adenocarcinoma; Stage IIIA Esophageal Adenocarcinoma; Stage IIIB Esophageal Adenocarcinoma; Stage IIIC Esophageal Adenocarcinoma
MeSH Terms: conditions — Adenocarcinoma Of Esophagus | interventions — Paclitaxel; Taxes; Carboplatin; Oxaliplatin; Leucovorin; Fluorouracil; Radiotherapy; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm I (paclitaxel, carboplatin, radiation therapy, surgery) (Experimental): INDUCTION: Patients receive chemotherapy with carboplatin and paclitaxel. Patients receive carboplatin (AUC=2) and paclitaxel (90 mg/m2) intravenously on days 1 and 8 of a 21 day treatment cycle for two cycles (total of 6 weeks).
  CHEMORADIATION THERAPY: Patients receive carboplatin (AUC=2) and paclitaxel (50 mg/m2) intravenously once weekly for five weeks throughout the duration of their radiation which is daily (Monday through Friday).
  SURGERY: Approximately 4-10 weeks after completion of chemoradiation therapy, patients undergo esophagectomy at the discretion of the treating team.
  Interventions: Drug: Paclitaxel; Drug: Carboplatin; Radiation: Radiation Therapy; Procedure: Therapeutic Conventional Surgery; Other: Laboratory Biomarker Analysis
- Arm II (combination chemotherapy, radiation therapy, surgery) (Experimental): INDUCTION: Patients receive mFOLFOX6 where they get oxaliplatin 85 mg/m2 intravenously on day 1, leucovorin 400 mg/m2 IV on day 1, 5-FU 400 mg/m2 IV on day 1 and then 5FU at 2400 mg/m2 IV to be administered over a 46 hour period. This is repeated every 2 weeks for 3 cycles (total of 6 weeks).
  CHEMORADIATION THERAPY: Patients receive oxaliplatin 85 mg/m2 IV on day 1 every 2 weeks for a total of 3 cycles (6 weeks) as well as 5FU 300 mg/m2/day over 96 hours via continuous infusion each week of radiation for a total of 6 weeks.
  SURGERY: Approximately 4-10 weeks after completion of chemoradiation therapy, patients undergo esophagectomy at the discretion of the treating team.
  Interventions: Drug: Oxaliplatin; Drug: Leucovorin Calcium; Drug: Fluorouracil; Radiation: Radiation Therapy; Procedure: Therapeutic Conventional Surgery; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Drug: Paclitaxel — Given IV or IVPB
  Other Names: Anzatax; TAX
  Arms: Arm I (paclitaxel, carboplatin, radiation therapy, surgery)
Drug: Carboplatin — Given IV or IVPB
  Arms: Arm I (paclitaxel, carboplatin, radiation therapy, surgery)
Drug: Oxaliplatin — Given IV
  Arms: Arm II (combination chemotherapy, radiation therapy, surgery)
Drug: Leucovorin Calcium — Given IV
  Other Names: CF
  Arms: Arm II (combination chemotherapy, radiation therapy, surgery)
Drug: Fluorouracil — Given IV
  Arms: Arm II (combination chemotherapy, radiation therapy, surgery)
Radiation: Radiation Therapy — Undergo radiation therapy
  Other Names: Cancer Radiotherapy; Irradiate; Irradiated; Irradiation; RT
Procedure: Therapeutic Conventional Surgery — Undergo esophagectomy
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This randomized pilot phase II trial studies how well molecular phenotyping works in predicting response in patients with stage IB-III esophageal cancer who are receiving carboplatin and paclitaxel or oxaliplatin, leucovorin calcium, and fluorouracil. Studying the genes in a patients tumor cells before and after chemotherapy may help in understanding if there are specific features of the tumor cells that make a person more or less likely to respond to treatment and how these features may be affected by treatment.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate gene and micro ribonucleic acid (miRNA) expression levels in patients with esophageal adenocarcinoma prior to receiving chemotherapy and identify relative expression differences between patients responding and not responding to treatment with carboplatin and paclitaxel or 5-fluorouracil (fluorouracil) and oxaliplatin as measured by fluorodeoxyglucose F-18 ([18F] FDG)-positron emission tomography (PET).

SECONDARY OBJECTIVES:

I. To evaluate the impact of treatment on expression patterns of both genes and miRNAs in patients with esophageal adenocarcinoma following treatment with either carboplatin and paclitaxel or 5-fluorouracil and oxaliplatin, and identify expression patterns associated with treatment response and resistance as assessed by (18F) FDG-PET.

II. To evaluate the expression patterns of genes and miRNAs in patients with esophageal adenocarcinoma prior to and following a full neoadjuvant combined-modality treatment program with either carboplatin and paclitaxel or 5-fluorouracil and oxaliplatin chemotherapy plus radiation, and identify relative expression differences between patients achieving a pathologic complete response and patients not achieving a pathologic complete response.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I:

INDUCTION: Patients receive carboplatin (IV) and paclitaxel intravenously (IV) on days 1 and 8 of a 21 day cycle for two cycles (total of 6 weeks).

CHEMORADIATION THERAPY: Patients receive carboplatin (AUC=2) and paclitaxel (50 mg/m2) intravenously once weekly for five weeks throughout the duration of their radiation which is daily (Monday through Friday). This will be given in combination with radiation therapy to a total of 50.4Gy using 180cGy fractions.

ARM II:

INDUCTION: Patients receive mFOLFOX6 where they get oxaliplatin 85 mg/m2 intravenously on day 1, leucovorin 400 mg/m2 IV on day 1, 5-FU 400 mg/m2 IV on day 1 and then 5FU at 2400 mg/m2 IV to be administered over a 46 hour period. This is repeated every 2 weeks for 3 cycles (total of 6 weeks).

CHEMORADIATION THERAPY: Patients receive chemoradiation with oxaliplatin 85 mg/m2 IV on day 1 every 2 weeks for a total of 3 cycles (6 weeks) as well as 5FU 300 mg/m2/day over 96 hours via continuous infusion each week of radiation for a total of 6 weeks. This will be given in combination with radiation therapy to a total of 50.4Gy using 180cGy fractions.

SURGERY: In both arms, approximately 4-10 weeks after completion of chemoradiation therapy, patients undergo esophagectomy at the discretion of the treating team.

After completion of study treatment, patients are followed up at 30 days and then periodically thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed localized (T1N1-3M0 or T2-4NanyM0, stage IB-III) Siewert type 1 or type 2 esophageal adenocarcinoma that is amenable to surgical resection as determined by a thoracic surgeon and for which all disease (primary tumor and involved lymph nodes) can be treated with radiation, as determined by a radiation oncologist
* Patients may not have received any prior chemotherapy, biologic therapy or radiation therapy for management of their disease; chemotherapy or biologic therapy administered for treatment of another primary malignancy are permitted if treatment was greater than 5 years ago
* Patients must have an Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* Patients must have a life expectancy of > 3 months, in the opinion of and as documented by the investigator
* Hemoglobin >= 10.0 g/dl
* Absolute neutrophil count >= 1,500/mcL
* Platelet count >= 100,000/mcL
* Total bilirubin within normal institutional limits
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) =< 2.5 X institutional upper limit of normal
* Alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 X institutional upper limit of normal
* Serum creatinine within normal institutional limits OR creatinine clearance >= 60 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal (as calculated by Cockcroft-Gault)
* Patients must have an avid primary tumor with an standardized uptake value (SUV) of >= 5 on baseline (18F) FDG-PET/computed tomography (CT) imaging
* Men must agree to use adequate contraception (double barrier method of birth control or abstinence) 1 week prior to study entry, for the duration of study participation and for 1 month after completing combined modality treatment with chemotherapy and radiation; should a male patient's female partner become pregnant or suspect that she is pregnant while her partner is participating in this study, the treating physician should be informed immediately
* Patients must have the ability to understand and the willingness to sign a written informed consent document
* This study will be limited to enrollment of Caucasian males only

Exclusion Criteria:

* Patients who are receiving any chemotherapy, biologic therapy, radiation therapy or any investigational agent
* Patients with metastatic disease
* Patients with a history of allergic reactions attributed to compounds of similar chemical or biologic composition to platinums, taxanes or fluoropyrimidines
* Patients who have previously received radiation therapy to the chest or abdomen such that there would be overlap between the previous and current radiation field
* Patients with uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Patients with human immunodeficiency virus (HIV) whom are not receiving antiretroviral therapy
* Patients with another malignancy within the past 5 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2015-02; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Eads, Principal Investigator — Case Comprehensive Cancer Center
Locations (1):
- Case Comprehensive Cancer Center, Cleveland, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm I (Paclitaxel, Carboplatin, Radiation Therapy, Surgery) | Arm II (Combination Chemotherapy, Radiation Therapy, Surgery)
Started | 0 | 1
Completed | 0 | 0
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: Number of patients initially enrolled on study. 0 patients completed the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Paclitaxel, Carboplatin, Radiation Therapy, Surgery) | Arm II (Combination Chemotherapy, Radiation Therapy, Surgery) | Total
Number analyzed (Participants) | 0 | 1 | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 1 | 1
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 1 | 1
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States |  | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Relative Expression Differences in Individual Genes and Gene Profiles Between Patients Responding and Not Responding to Treatment, as Assessed by (18F) FDG-PET
Description: Baseline gene profiles will be compared for 10 (18F) FDG-PET responders vs. 15 (18F) FDG-PET non-responders per treatment regimen using a t-test and p-values will be corrected for multiple comparisons by calculating the false discovery rate (FDR) p-value (filtering on a FDR p-value < 0.05). Top genes identified will be tested in combination for their sensitivity and specificity using logistic regression models.
Time Frame: Baseline
Population: No patients completed study and no patients were enrolled on the comparison group arm. No analysis could be completed.
Arm/Group | Arm I (Paclitaxel, Carboplatin, Radiation Therapy, Surgery) | Arm II (Combination Chemotherapy, Radiation Therapy, Surgery)
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Relative Expression Differences in Individual microRNAs and microRNA Profiles Between Patients Responding and Not Responding to Treatment, Assessed by (18F) FDG-PET
Description: Baseline microRNA profiles will be compared for 10 (18F) FDG-PET responders vs. 15 (18F) FDG-PET non-responders per treatment regimen using a t-test and p-values will be corrected for multiple comparisons by calculating the FDR p-value (filtering on a FDR p-value < 0.05). Top microRNAs identified will be tested in combination for their sensitivity and specificity using logistic regression models.
Time Frame: Baseline
Population: No patients completed study and no patients were enrolled on the comparison group arm. No analysis could be completed.
Arm/Group | Arm I (Paclitaxel, Carboplatin, Radiation Therapy, Surgery) | Arm II (Combination Chemotherapy, Radiation Therapy, Surgery)
Number analyzed (Participants) | 0 | 0

3. Primary Outcome: Biological Pathway Perturbation Upon Exposure to Chemotherapy
Description: Predefined signatures of biological pathway activities will be evaluated in order to identify pathway perturbation upon exposure to chemotherapy. Significant pathway modulations upon brief exposure will then be evaluated for association with clinical response using non-parametric tests such as the Wilcoxon signed-rank test. In all cases, statistical correction to account for multiple hypothesis testing will be employed and pathways with a false discovery rate of 10% or lower will be considered as significant.
Time Frame: Up to 6 weeks
Population: No patients completed study and no patients were enrolled on the comparison group arm. No analysis could be completed.
Arm/Group | Arm I (Paclitaxel, Carboplatin, Radiation Therapy, Surgery) | Arm II (Combination Chemotherapy, Radiation Therapy, Surgery)
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Relative Expression Differences Between Baseline and Post-induction Chemotherapy Specimens of Individual Genes and Gene Expression Profiles
Description: Changes in baseline and post-treatment gene expression levels will be calculated between (18F) FDG-PET responders and non-responders, filtering for expression level changes of >= 0.20. Differences in expression level change per treatment regimen will be calculated using a t-test and p-values will be corrected for multiple comparisons by calculating FDR p-value (filtering on a FDR p-value < 0.05). Top genes identified will be tested in combination for their sensitivity and specificity using logistic regression models to predict responsiveness or resistance to each individual treatment regimen.
Time Frame: Baseline to post-induction (36-43 days)
Population: No patients completed study and no patients were enrolled on the comparison group arm. No analysis could be completed.
Arm/Group | Arm I (Paclitaxel, Carboplatin, Radiation Therapy, Surgery) | Arm II (Combination Chemotherapy, Radiation Therapy, Surgery)
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Relative Expression Differences Between Baseline and Post-induction Chemotherapy Specimens of Individual microRNAs and microRNA Profiles
Description: Changes in baseline and post-treatment microRNA levels will be calculated between (18F) FDG-PET responders and non-responders, filtering for expression level changes of >= 0.20. Differences in expression level change per treatment regimen will be calculated using a t-test and p-values will be corrected for multiple comparisons by calculating FDR p-value (filtering on a FDR p-value < 0.05). Top microRNAs identified will be tested in combination for their sensitivity and specificity using logistic regression models to predict responsiveness or resistance to each individual treatment regimen.
Time Frame: Baseline to post-induction (36-43 days)
Population: No patients completed study and no patients were enrolled on the comparison group arm. No analysis could be completed.
Groups:
- Arm I (Paclitaxel, Carboplatin, Radiation Therapy, Surgery): Experimental: Arm I (paclitaxel, carboplatin, radiation therapy, surgery) INDUCTION: Patients receive chemotherapy with carboplatin and paclitaxel. Patients receive carboplatin (AUC=2) and paclitaxel (90 mg/m2) intravenously on days 1 and 8 of a 21 day treatment cycle for two cycles (total of 6 weeks).
  CHEMORADIATION THERAPY: Patients receive carboplatin (AUC=2) and paclitaxel (50 mg/m2) intravenously once weekly for five weeks throughout the duration of their radiation which is daily (Monday through Friday).
  SURGERY: Approximately 4-10 weeks after completion of chemoradiation therapy, patients undergo esophagectomy at the discretion of the treating team.
Arm/Group | Arm I (Paclitaxel, Carboplatin, Radiation Therapy, Surgery) | Arm II (Combination Chemotherapy, Radiation Therapy, Surgery)
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Relative Expression Differences in Baseline Individual Genes and Gene Expression Profiles Between Patients Achieving and Not Achieving a Pathologic Complete Response Following Treatment
Description: Baseline gene expression profiles for 8 pathologic complete responders vs. 17 patients not achieving a pathologic complete response per treatment regimen using a t-test will be compared. Top genes will be tested in combination for their sensitivity and specificity using logistic regression models to predict achievement of a pathologic complete response vs. patients not achieving a pathologic complete response.
Time Frame: Baseline
Population: No patients completed study and no patients were enrolled on the comparison group arm. No analysis could be completed.
Groups:
- Arm I (Paclitaxel, Carboplatin, Radiation Therapy, Surgery): INDUCTION:Patients receive chemotherapy with carboplatin and paclitaxel. Patients receive carboplatin (AUC=2) and paclitaxel (90 mg/m2) intravenously on days 1 and 8 of a 21 day treatment cycle for two cycles (total of 6 weeks).
  CHEMORADIATION THERAPY: Patients receive carboplatin (AUC=2) and paclitaxel (50 mg/m2) intravenously once weekly for five weeks throughout the duration of their radiation which is daily (Monday through Friday).
  SURGERY: Approximately 4-10 weeks after completion of chemoradiation therapy, patients undergo esophagectomy at the discretion of the treating team.
Arm/Group | Arm I (Paclitaxel, Carboplatin, Radiation Therapy, Surgery) | Arm II (Combination Chemotherapy, Radiation Therapy, Surgery)
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Relative Expression Differences in Baseline Individual microRNAs and microRNA Profiles Between Patients Achieving and Not Achieving a Pathologic Complete Response Following Treatment
Description: Baseline microRNA profiles for 8 pathologic complete responders vs. 17 patients not achieving a pathologic complete response per treatment regimen using a t-test will be compared. Top microRNAs will be tested in combination for their sensitivity and specificity using logistic regression models to predict achievement of a pathologic complete response vs. patients not achieving a pathologic complete response.
Time Frame: Baseline
Population: No patients completed study and no patients were enrolled on the comparison group arm. No analysis could be completed.
Arm/Group | Arm I (Paclitaxel, Carboplatin, Radiation Therapy, Surgery) | Arm II (Combination Chemotherapy, Radiation Therapy, Surgery)
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Relative Expression Differences Between Baseline and Post-induction Gene Expression Levels/Profiles Between Patients Achieving and Not Achieving a Pathologic Complete Response Following Treatment
Description: Changes in baseline and post-treatment gene expression level/profiles will be compared between 8 pathologic responders vs. 17 patients not achieving a pathologic complete response per treatment regimen, filtering for expression levels changes of 0.20 and above. Differences in expression level changes per treatment regimen will be calculated using a t-test. Top genes will be tested in combination for their sensitivity and specificity using logistic regression models to predict achievement of a pathologic complete response vs. patients not achieving a pathologic complete response.
Time Frame: Baseline to post-induction (36-43 days)
Population: No patients completed study and no patients were enrolled on the comparison group arm. No analysis could be completed.
Arm/Group | Arm I (Paclitaxel, Carboplatin, Radiation Therapy, Surgery) | Arm II (Combination Chemotherapy, Radiation Therapy, Surgery)
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Relative Expression Differences Between Baseline and Post-induction microRNA Levels/Profiles Between Patients Achieving and Not Achieving a Pathologic Complete Response Following Treatment
Description: Changes in baseline and post-treatment microRNA level/profiles will be compared between 8 pathologic responders vs. 17 patients not achieving a pathologic complete response per treatment regimen, filtering for expression levels changes of 0.20 and above. Differences in expression level changes per treatment regimen will be calculated using a t-test. Top microRNAs will be tested in combination for their sensitivity and specificity using logistic regression models to predict achievement of a pathologic complete response vs. patients not achieving a pathologic complete response.
Time Frame: Baseline to post-induction (36-43 days)
Population: No patients completed study and no patients were enrolled on the comparison group arm. No analysis could be completed.
Arm/Group | Arm I (Paclitaxel, Carboplatin, Radiation Therapy, Surgery) | Arm II (Combination Chemotherapy, Radiation Therapy, Surgery)
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Occurrence of Grade 3 or 4 Toxicity Per the National Cancer Institute Common Toxicity Criteria for Adverse Events (NCI CTCAE) Version 4.0
Description: Toxicities will be summarized as the percentage of patients experiencing each type and grade of event according to treatment group. Patients who receive at least one dose of treatment will be included in the analysis.
Time Frame: Up to 30 days after the end of treatment
Population: No patients completed study and no patients were enrolled on the comparison group arm. No analysis could be completed.
Arm/Group | Arm I (Paclitaxel, Carboplatin, Radiation Therapy, Surgery) | Arm II (Combination Chemotherapy, Radiation Therapy, Surgery)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Groups:
- Arm I (Paclitaxel, Carboplatin, Radiation Therapy, Surgery): INDUCTION: Patients receive paclitaxel IV over 60 minutes and carboplatin intravenously IV over 30 minutes on days 1 and 8. Treatment repeats every 21 days for 2 courses in the absence of disease progression or unacceptable toxicity.
  CHEMORADIATION THERAPY: Patients receive paclitaxel IVPB over 60 minutes and carboplatin IVPB over 30 minutes on days 8 and 22. Patients also undergo radiation therapy QD 5 days a week. Treatment continues for 5-6 weeks in the absence of disease progression or unacceptable toxicity.
  SURGERY: Approximately 4-10 weeks after completion of chemoradiation therapy, patients undergo esophagectomy at the discretion of the treating team.
  Paclitaxel: Given IV or IVPB
  Carboplatin: Given IV or IVPB
  Radiation Therapy: Undergo radiation therapy
  Therapeutic Conventional Surgery: Undergo esophagectomy
  Laboratory Biomarker Analysis: Correlative studies
- Arm II (Combination Chemotherapy, Radiation Therapy, Surgery): INDUCTION: Patients receive oxaliplatin IV over 2-6 hours, leucovorin calcium IV over 2 hours, and fluorouracil IV continuously over 46-48 hours. Treatment repeats every 14 days for 3 courses in the absence of disease progression or unacceptable toxicity.
  CHEMORADIATION THERAPY: Patients receive oxaliplatin IV over 2-6 hours on days 1, 15, and 29 and fluorouracil IV continuously over 96 hours on days 1, 8, 15, 22, and 29. Patients also undergo radiation therapy QD 5 days a week for 5-6 weeks. Treatment continues in the absence of disease progression or unacceptable toxicity.
  SURGERY: Approximately 4-10 weeks after completion of chemoradiation therapy, patients undergo esophagectomy at the discretion of the treating team.
  Oxaliplatin: Given IV
  Leucovorin Calcium: Given IV
  Fluorouracil: Given IV
  Radiation Therapy: Undergo radiation therapy
  Therapeutic Conventional Surgery: Undergo esophagectomy
  Laboratory Biomarker Analysis: Correlative studies
Arm/Group | Arm I (Paclitaxel, Carboplatin, Radiation Therapy, Surgery) | Arm II (Combination Chemotherapy, Radiation Therapy, Surgery)
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/1
Other Adverse Events (participants affected / at risk) | 0/0 | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes